CLINICAL TRIAL: NCT00191880
Title: A Phase IIIb Open-Label Trial of Atomoxetine Hydrochloride to Evaluate Academic Outcome in Children Ages 8 to 11 Years With Attention-Deficit/Hyperactivity Disorder
Brief Title: Open-Label Trial of Atomoxetine to Evaluate Academic Outcome in Children Ages 8-11 Years With Attention Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7649; B4Z-CA-LYCS
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: atomoxetine

SUMMARY:
Open-label trial of Atomoxetine to Evaluate Academic Outcome in Children Ages 8-11 years with Attention- Deficit/Hyperactivity Disorder

ELIGIBILITY:
Inclusion Criteria:

-Patients must have ADHD, be psychotropic medication naive and be outpatients who are at least 8 years of age and not more than 10 years of age at Visit 1 (that is, not yet reached their 11 birthday) so that all year testing will be completed before the child reaches age 12.

Exclusion Criteria:

-Patients with current or past history of Bipolar I or II disorder, psychosis, autism, Asperger's syndrome, pervasive developmental disorder, conduct disorder, seizure disorder or serious suicidal risk are excluded

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2004-05; Study Completion 2006-06

PRIMARY OUTCOMES:
The primary objective of this study is to assess the correlation of change from baseline to one year in ADHD symptoms as measured by the Attention Deficit/Hyperactivity Disorder Rating Scale- IV-
Parent Version: Investigator Administered and Scored,
total score, with change from baseline in academic achievement of medication-naive patients treated with atomoxetine at one year as measured by the total
of the composite scores of the broad reading, broad math, and broad language subtests of the Woodcock-Johnson Tests of Achievement (WJII)

SECONDARY OUTCOMES:
To Assess the correlation of change from baseline to one year or at study discontinuation in ADHD symptoms as measured by the ADHDRS-IV-Parent:Inv with change from baseline with each of the academic achievement composite scores of the broad reading, broa

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- Canada (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Calgary
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Edmonton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Montreal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saskatoon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Scarborough
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, St. Johns
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Toronto

REFERENCES:
- [Derived] Dickson RA, Maki E, Gibbins C, Gutkin SW, Turgay A, Weiss MD. Time courses of improvement and symptom remission in children treated with atomoxetine for attention-deficit/hyperactivity disorder: analysis of Canadian open-label studies. Child Adolesc Psychiatry Ment Health. 2011 May 11;5:14. doi: 10.1186/1753-2000-5-14. PMID 21569378